CLINICAL TRIAL: NCT01696942
Title: Use of Certolizumab Following Ileocolectomy Lowers Endoscopic and Histological Recurrence Rates for Crohn's Disease at One Year Compared to Mesalamine
Brief Title: Cimzia Versus Mesalamine for Crohn's Recurrence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, David B. Stewart, MD, FACS, FASCRS, Assistant Professor of Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36497
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Results first posted 2017-10-10 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; certolizumab; mesalamine; recurrence
MeSH Terms: conditions — Crohn Disease; Recurrence | interventions — Certolizumab Pegol; Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cimzia treatment arm (Experimental): Beginning at 4 weeks after surgery, patients would be randomly assigned using a pulled card method to receive certolizumab at a dose of 400 mg subcutaneously at weeks 4, 6, and 8 after surgery, and then every 4 weeks thereafter up to 12 months after enrollment.
  Interventions: Drug: Cimzia
- Mesalamine treatment arm (Active Comparator): Beginning at 4 weeks after surgery, patients would be randomly assigned to receive mesalamine 800 mg orally three times daily for twelve months following enrollment.
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Cimzia — 400 mg subcutaneously at weeks 4, 6, and 8 after surgery, and then every 4 weeks
  Other Names: Certolizumab
  Arms: Cimzia treatment arm
Drug: Mesalamine — mesalamine 800 mg orally three times daily
  Arms: Mesalamine treatment arm

SUMMARY:
Hypothesis: Cimzia provides superior reduction in endoscopic and clinical recurrence rates compared to mesalamine in the treatment of Crohn's disease one-year following ileocolectomy for Crohn's disease.

1. To evaluate the difference in clinical recurrence rates between certolizumab and mesalamine after 4 weeks, 3 months, 6 months, 9 months, and 12 months of use following ileocolectomy for Crohn's disease using the Crohn's Disease Activity Index (CDAI).
2. To compare the endoscopic recurrence rates at one year following surgery between patients treated with certolizumab and mesalamine.
3. To compare medication side-effects and tolerance of therapy, including the need to interrupt therapy due to side-effects, the incidence of opportunistic infections, and a general assessment of each patient's health and well-being using the short-form 36 (SF-36).

DETAILED DESCRIPTION:
Crohn's disease is an autoimmune, pan-intestinal disease which can affect any portion of the alimentary tract, but which has a preference for the small intestine, the colon, and the anus. It is now well established that Crohn's disease most commonly presents with an ileocolic distribution, followed by involvement of the small intestine, the colon, and the anus. Treatment for Crohn's disease is principally medical, reserving surgery to address complications from the disease which cannot be adequately resolved with medication alone. The single greatest challenge in treating this incurable disease is dealing with its recurrence rate. The cumulative probability of disease recurrence is quite high, with 75% of Crohn's patients requiring abdominal surgery at some point during their life.

Following surgery, recurrence rates are significant, varying depending on the manner in which recurrence is defined. With regard to clinical recurrences, where the recrudescence of the disease is associated with symptoms caused by new intestinal lesions, the recurrence rate is 10-20% per year.In some instances, clinical recurrences can appear within 3 months of surgery. Taking into account the need for additional surgery as defining a "surgical recurrence", reoperation rates for Crohn's disease range from 16% to 65% 10 years after a previous surgery. When recurrence is viewed from the vantage point of evidence of new Crohn's disease activity based on radiographic studies, radiographic recurrences range from 41-60% over the first 10 years following surgery. One of the most common measures of recurrence has become demonstrating evidence of new Crohn's disease activity based on colonoscopy. This endoscopic recurrence has consistently been shown to be as high as 50-75% at 3 months after surgery, and 50-90% at 12 months. It is widely accepted by physicians treating Crohn's patients that the appearance of endoscopic lesions has prognostic significance, as endoscopic evidence of Crohn's disease temporally precedes radiographic, clinical and surgical recurrences.

The role that Cimzia should play in preventing recurrence of Crohn's disease following ileocolectomy for Crohn's disease remains to be determined, as does its relative advantages and disadvantages compared to the use of mesalamine.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age or older with Crohn's disease of any phenotype (luminal disease, perforating disease, stricturing disease) with an ileocolic distribution.
* Ileocolic Crohn's disease severe enough to require ileocolectomy (either open or laparoscopic).

Exclusion Criteria:

* Patients younger than 18 years of age, as there is little data on pediatric patients and since the Colorectal Surgery service only treats patients 18 years of age or older.
* Patients undergoing an ileocolectomy for any reason besides Crohn's disease.
* Patients requiring a stoma.
* Patients with short-bowel syndrome.
* Patients who are incarcerated, due to difficulties with frequent clinic visits given their incarceration and transportation issues.
* Patients who received previous anti-TNF therapy from infliximab or adalimumab within three months of surgery, or patients who have a history of a severe hypersensitivity reaction to infliximab or adalimumab
* Patients with a positive PPD and a suspicious finding on a chest x-ray suggestive of tuberculosis, or any patient with a history of tuberculosis.
* Patients who require postoperative therapy besides either mesalamine or certolizumab (steroids, antibiotics, and immunomodulator therapy would not be permitted starting at 4 weeks after ileocolectomy).
* Patients with significant psychiatric disorders (i.e. schizophrenia) and those with significant cognitive disorders, due to the difficulties with this patient group remaining compliant with frequent clinic visits, and due to the difficulty evaluating quality of life measures in these patients.
* Patients with a history of malignancy.
* Patients with a history of any demyelinating neurologic disease or a history of seizures.
* Patients with a history of severe congestive heart failure.
* Patients with a history of hepatitis B or C virus.
* Patients who are pregnant or who become pregnant.
* Involvement in any other clinical studies which use study medications.
* The subject has a condition, which, in the opinion of the investigator, would compromise the study or well-being of the subject or prevent the subject from meeting or performing the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Stewart, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Whelan G, Farmer RG, Fazio VW, Goormastic M. Recurrence after surgery in Crohn's disease. Relationship to location of disease (clinical pattern) and surgical indication. Gastroenterology. 1985 Jun;88(6):1826-33. doi: 10.1016/0016-5085(85)90007-1. PMID 3996839
- [Background] Mekhjian HS, Switz DM, Watts HD, Deren JJ, Katon RM, Beman FM. National Cooperative Crohn's Disease Study: factors determining recurrence of Crohn's disease after surgery. Gastroenterology. 1979 Oct;77(4 Pt 2):907-13. No abstract available. PMID 467942
- [Background] Kyle J. Prognosis after ileal resection for Crohn's disease. Br J Surg. 1971 Oct;58(10):735-7. doi: 10.1002/bjs.1800581006. No abstract available. PMID 5097949
- [Background] Lennard-Jones JE, Stalder GA. Prognosis after resection of chronic regional ileitis. Gut. 1967 Aug;8(4):332-6. doi: 10.1136/gut.8.4.332. No abstract available. PMID 6039720
- [Background] Greenstein AJ, Sachar DB, Pasternack BS, Janowitz HD. Reoperation and recurrence in Crohn's colitis and ileocolitis; Crude and cumulative rates. N Engl J Med. 1975 Oct 2;293(14):685-90. doi: 10.1056/NEJM197510022931403. PMID 1160935
- [Background] Regueiro M, Schraut W, Baidoo L, Kip KE, Sepulveda AR, Pesci M, Harrison J, Plevy SE. Infliximab prevents Crohn's disease recurrence after ileal resection. Gastroenterology. 2009 Feb;136(2):441-50.e1; quiz 716. doi: 10.1053/j.gastro.2008.10.051. Epub 2008 Oct 31. PMID 19109962
- [Background] Cottone M, Mocciaro F, Orlando A. Infliximab prevents Crohn's disease recurrence after ileal resection. Expert Rev Gastroenterol Hepatol. 2009 Jun;3(3):231-4. doi: 10.1586/egh.09.13. No abstract available. PMID 19485805
- [Background] Schreiber S. Certolizumab pegol for the treatment of Crohn's disease. Therap Adv Gastroenterol. 2011 Nov;4(6):375-89. doi: 10.1177/1756283X11413315. PMID 22043230
- [Background] Sandborn WJ, Schreiber S, Feagan BG, Rutgeerts P, Younes ZH, Bloomfield R, Coteur G, Guzman JP, D'Haens GR. Certolizumab pegol for active Crohn's disease: a placebo-controlled, randomized trial. Clin Gastroenterol Hepatol. 2011 Aug;9(8):670-678.e3. doi: 10.1016/j.cgh.2011.04.031. Epub 2011 May 13. PMID 21642014
- [Background] Feagan BG, Sandborn WJ, Wolf DC, Coteur G, Purcaru O, Brabant Y, Rutgeerts PJ. Randomised clinical trial: improvement in health outcomes with certolizumab pegol in patients with active Crohn's disease with prior loss of response to infliximab. Aliment Pharmacol Ther. 2011 Mar;33(5):541-50. doi: 10.1111/j.1365-2036.2010.04568.x. Epub 2011 Jan 12. PMID 21223344

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cimzia Treatment Arm | Mesalamine Treatment Arm
Started | 5 | 5
Completed | 3 | 2
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — screen failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cimzia Treatment Arm | Mesalamine Treatment Arm | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Recurrence Rates of Crohn's Disease
Description: To evaluate the difference in clinical recurrence rates between certolizumab and mesalamine after 4 weeks, 3 months, 6 months, 9 months, and 12 months of use following ileocolectomy for Crohn's disease using the Crohn's Disease Activity Index (CDAI). CDAI scores of 150 or greater are considered a recurrence.
Time Frame: 4 weeks, 3 months, 6 months, 9 months, and 12 months
Population: Subjects who received CDAI questionnaire. Number of participants fluctuates due to withdrawals and missed appointments.
Measure: Count of Participants; unit: Participants
Arm/Group | Cimzia Treatment Arm | Mesalamine Treatment Arm
Number analyzed (Participants) | 5 | 3
Participants
  4 week CDAI recurrence | 3 | 1
  3 month CDAI reccurence: number analyzed (Participants) | 4 | 3
  3 month CDAI reccurence | 2 | 1
  6 month CDAI recurrence: number analyzed (Participants) | 3 | 3
  6 month CDAI recurrence | 1 | 2
  9 month CDAI recurrence: number analyzed (Participants) | 3 | 2
  9 month CDAI recurrence | 2 | 0
  12 month CDAI recurrence: number analyzed (Participants) | 2 | 2
  12 month CDAI recurrence | 0 | 0

2. Secondary Outcome: Number of Participants With Endoscopic Recurrence of Crohn's Disease
Description: To compare the endoscopic recurrence rates at one year following surgery between patients treated with certolizumab and mesalamine.
Time Frame: One year following enrollment
Population: Subjects available for colonoscopy at 12 month visit. This visit was sometimes separated from the overall 12-month visit so only 1 (cimzia) and 2 (mesalamine) patients respectively had the colonoscopy performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cimzia Treatment Arm | Mesalamine Treatment Arm
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cimzia Treatment Arm | Mesalamine Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimzia Treatment Arm (N=5) | Mesalamine Treatment Arm (N=5)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
dehydration (General disorders) | 1 (1) | 1 (1)
Episcleritis (Eye disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (2) | 1 (1)
Abdominal Pain (General disorders) | 2 (2) | 0 (0)
Perianal rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
papular rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal ache (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ulcer (anastamotic) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Attention Deficit (Psychiatric disorders) | 1 (1) | 0 (0)
melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (2)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
fecal calprotectin elevation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1)
Elevated CRP (General disorders) | 1 (1) | 0 (0)
colon inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
cramping with BM (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's flare (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No